CLINICAL TRIAL: NCT05975827
Title: Sterile Wound Care Liquid Dressing in Treatment of Diabetic Ulcer in Necrosis Stable Stage: a Randomized Control Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Long2024-DFU-Sterile dressing
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Ulcers; Diabetic Ulcers in Necrosis Stable Stage
Keywords: Diabetic Ulcers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterile Wound Care Liquid Dressing (Experimental)
  Interventions: Device: Sterile Wound Care Liquid Dressing
- Control (No Intervention)

INTERVENTIONS:
Device: Sterile Wound Care Liquid Dressing — Sterile wound care liquid dressing is used in the wound treatment
  Arms: Sterile Wound Care Liquid Dressing

SUMMARY:
This study aimed to investigate methods for promoting infection control, reducing tissue edema, and preventing excessive spread in diabetes foot ulcers in the necrosis stable stage. Additionally, it sought to explore potential indications for the use of aseptic wound care liquid dressings in these ulcers, with the goal of obtaining evidence-based medical data on their clinical efficacy.

Participants will be assigned with a 1:1 ratio into intervention group and control group.

Participants in the intervention group will be irrigated with sterile liquid dressing for each wound treatment on the basis of clinical standard treatment protocols for 2 weeks, until the end of the 2-week observation period. Participants in the control group will be irrigated with normal saline for each wound treatment for 2 weeks on the basis of the clinical standard diagnosis and treatment plan, until the end of the 2-week observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Severe diseases such as acute myocardial infarction, heart failure, hepatitis, shock, respiratory failure, renal failure etc., which have not been corrected.
2. Poor glycemic control; fasting blood glucose >15mmol/L; glycosylated hemoglobin >12%.
3. Active bleeding within the wound that prevents implementation of standard basic treatment protocols.
4. Serum albumin <20g/L; hemoglobin <60g/L; platelets <50×10^9/L
5. Advanced malignant tumor patients
6. Autoimmune disease activity period
7. History of allergy to aseptic wound care liquid dressing
8. Patient unable to cooperate or has mental disorders
9. Pregnant and lactating women
10. Eye injuries and natural cavities such as ear canal, nasal cavity or abdominal cavity
11. Skin tumors
12. Active skin diseases
13. According to the researcher's judgment, patients who clearly have factors affecting wound healing that cannot be removed are not suitable for this study or cannot comply with the requirements of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
2-week reduction rate of wound area | 2-week

SECONDARY OUTCOMES:
2-week wound healing rate | 2-week